CLINICAL TRIAL: NCT06985420
Title: The Impact of the Menstrual Cycle on Innate Immune Cell Activation, Recruitment, and Adhesion Dynamics During Recovery From Damaging Resistance Exercise: Role of Neutrophils and Systemic Chemokines.
Brief Title: The Effect of the Menstrual Cycle on Immune Cell Activity and Recovery After Resistance Exercise
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Jessica Moon, Graduate Research Assistant, PhD Candidate, Principal Investigator, University of Central Florida
Other Study IDs: STUDY00006956
Record Dates: First submitted 2024-09-16; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Healthy Women; Menstruation; Resistance Exercise
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Resistance exercise — Resistance Exercise Protocols: Participants will perform exercises, including belt squats, hex bar deadlifts, and plyometric drop jumps. The load and intensity will be standardized based on each participant's 1-repetition maximum (1RM) to ensure uniformity across trials.
Other: Menstrual Cycle Phases — Menstrual Cycle Phases: The key exposure variable is the phase of the menstrual cycle, with participants being assessed during the early follicular, late follicular, and mid-luteal phases.

SUMMARY:
The goal of this observational study is to learn how the menstrual cycle affects immune cell activation, recruitment, and recovery responses after resistance exercise in healthy, resistance-trained women aged 18-40. The main questions it aims to answer are:

Does the menstrual cycle influence neutrophil recruitment and adhesion after resistance exercise? Does the menstrual cycle affect markers of muscle damage and functional recovery? Researchers will compare three menstrual phases (early follicular, late follicular, and mid-luteal) to see if immune responses and recovery outcomes differ across these phases.

Participants will:

Complete resistance exercise protocols across three different menstrual cycle phases.

Provide blood samples to assess immune cell activation and muscle damage markers.

Track sleep, mood, and recovery with questionnaires and wear an accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 40.
* Must weigh at least 110 pounds.
* Healthy as determined by medical history, physical activity readiness, and menstrual cycle questionnaires.
* Actively resistance training for at least 6 months (minimum of 3 resistance training sessions per week, with at least one lower body session).
* Pre-menopausal and have a regular menstrual cycle (eumenorrheic), with a clear start of menses (early follicular phase).
* Not currently pregnant or planning to become pregnant during the study.
* Have not used hormonal birth control or intrauterine devices in the past 3 months (or three full menstrual cycles).
* Able to recall approximate start dates of their last 6 menstrual cycles.
* Willing to follow study instructions, including avoiding exercise, alcohol, and caffeine before testing visits.
* Free from previous or current lower body injuries that could limit performance.
* Not regularly taking any medications that could interfere with the study.
* Determined to have a high likelihood of successful blood draws by a certified phlebotomist.

Exclusion Criteria:

* Do not give consent to participate.
* Have been determined unfit to participate based on medical or activity history (using health questionnaires).
* Currently take prescription or over-the-counter medication that could affect the study results.
* Have a chronic illness requiring medical care.
* Not currently resistance-trained (don't meet the exercise requirement).
* Pregnant or planning to become pregnant during the study.
* Do not have regular periods or have been diagnosed as amenorrhoeic (absence of menstruation).
* Currently taking any performance-enhancing drugs.
* Currently using hormonal birth control or intrauterine devices (IUDs), or have used them in the past three months (or three full menstrual cycles).
* Determined unlikely to have a successful blood draw by a trained phlebotomist.
* Weigh less than 110 pounds.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Participants will be recruited from the local community and university setting, specifically from the University of Central Florida and surrounding areas. The population will consist of healthy, resistance-trained women aged 18 to 40 who are physically active and meet the criteria for regular menstrual cycles. Participants will likely be university students, staff, or individuals involved in local fitness and sports communities, with a focus on those who are familiar with structured resistance training. Recruitment will aim to reflect a diverse range of backgrounds while ensuring participants meet the health and exercise requirements of the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Recruitment and Adhesion Dynamics | From enrollment, through study completion, an average of 4 months.
  Measure: Neutrophil cell index (impedance reflecting neutrophil migration) using Real-Time Cell Analysis (RTCA). Objective: To assess the differences in neutrophil recruitment and adhesion across menstrual cycle phases (early follicular, late follicular, and mid-luteal).
  Time Frame: Assessed at 2 time points (baseline and 4 hours post exercise) on 3 experimental trial days (1 per menstrual cycle; up to 4 cycles per participant, over approximately 16 weeks).
Systemic Concentrations of CXCL8 | From enrollment, through study completion, an average of 4 months.
  Measure: Plasma levels of CXCL8 (interleukin-8). Objective: To evaluate if menstrual cycle phases influence systemic chemokine levels in response to exercise.
  Time Frame: Collected at 2 time points (baseline and 4 hours post exercise) on 3 experimental trial days (1 per menstrual cycle; up to 4 cycles per participant, over approximately 16 weeks).
Muscle Function and Recovery- Active Range of Motion | From enrollment, through study completion, an average of 4 months.
  Measure: Changes in active range of motion (AROM). Objective: To examine the impact of the menstrual cycle on functional recovery following resistance exercise.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days (1 per menstrual cycle; up to 4 cycles per participant, over approximately 16 weeks).
Muscle Function and Recovery- Pain Pressure Threshold | From enrollment, through study completion, an average of 4 months.
  Measure: Changes in pain pressure threshold (PPT). Objective: To examine the impact of the menstrual cycle on functional recovery following resistance exercise.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days (1 per menstrual cycle; up to 4 cycles per participant, over approximately 16 weeks).
Muscle Function and Recovery - Countermovement Jump | From enrollment, through study completion, an average of 4 months.
  Measure: Changes in countermovement jump (CMJ) height. Objective: To examine the impact of the menstrual cycle on functional recovery following resistance exercise.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days (1 per menstrual cycle; up to 4 cycles per participant, over approximately 16 weeks).
Muscle Function and Recovery - Maximal Voluntary Isometric Contraction | From enrollment, through study completion, an average of 4 months.
  Measure: Changes in maximal voluntary isometric contraction (MVIC). Objective: To examine the impact of the menstrual cycle on functional recovery following resistance exercise.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days (1 per menstrual cycle; up to 4 cycles per participant, over approximately 16 weeks).

SECONDARY OUTCOMES:
Systemic Concentrations of Myoglobin | From enrollment, through study completion, an average of 4 months.
  Measure: Plasma levels of myoglobin (MYB). Objective: To determine how menstrual cycle phases affect muscle damage/inflammation markers after resistance exercise.
  Time Frame: Collected at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total).
Systemic Concentrations of Creatine kinase | From enrollment, through study completion, an average of 4 months.
  Measure: Plasma levels of creatine kinase (CK). Objective: To determine how menstrual cycle phases affect muscle damage/inflammation markers after resistance exercise.
  Time Frame: Collected at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total).
Systemic Concentrations of C-Reactive Protein | From enrollment, through study completion, an average of 4 months.
  Measure: Plasma levels of C-reactive protein (CRP). Objective: To determine how menstrual cycle phases affect muscle damage/inflammation markers after resistance exercise.
  Time Frame: Collected at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total).
Subjective Measures of Perceived Recovery | From enrollment, through study completion, an average of 4 months.
  Measure: Perceived Recovery Status Scale score. Objective: To assess perceived recovery and performance across menstrual cycle phases.
  Time Frame: Assessed at 5 time points (baseline, immediately post, 4 hours, 24 hours, and 48 hours post-exercise) on up to 3 experimental trial days (approximately 16 weeks total).
Subjective Measures of Perceived Recovery | From enrollment, through study completion, an average of 4 months.
  Measure: Visual Analog Scale (VAS) ratings for recovery. Objective: To assess perceived recovery across menstrual cycle phases.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on up to 4 experimental trial days per participant (approximately 16 weeks total).
Subjective Measures of Fatigue | From enrollment, through study completion, an average of 4 months.
  Measure: Visual Analog Scale (VAS) ratings for fatigue. Objective: To assess perceived fatigue across menstrual cycle phases.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total).
Subjective Measures of Soreness | From enrollment, through study completion, an average of 4 months.
  Measure: Visual Analog Scale (VAS) ratings for soreness. Objective: To assess perceived soreness across menstrual cycle phases.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total).
Subjective Sleep Quality | Time Frame: From enrollment, through study completion, an average of 4 months.
  Measure: Groningen Sleep Quality Questionnaire (GSQQ). Objective: To investigate whether menstrual cycle phases impact subjective sleep quality.
  Time Frame: Assessed at 3 time points (baseline, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total)
Subjective Sleep Quality | From enrollment, through study completion, an average of 4 months.
  Measure: Self-Assessment of Sleep Survey (SASS-Y). Objective: To investigate whether menstrual cycle phases impact subjective sleep quality.
  Time Frame: Assessed at 1 time point (baseline) on 3 experimental trial days per participant (approximately 16 weeks total)
Objective Sleep Quality | From enrollment, through study completion, an average of 4 months.
  Measure: Actigraph Accelerometer data. Objective: To investigate whether menstrual cycle phases impact objective sleep quality.
  Time Frame: Continuously monitored from 72 hours before to 48 hours after exercise on each of 3 experimental trial days (approximately 16 weeks total).
Mood | From enrollment, through study completion, an average of 4 months.
  Measure: Profile of Mood States (POMS). Objective: To examine the influence of the menstrual cycle on mood during recovery from exercise.
  Time Frame: Assessed at 5 time points (baseline, immediately post-exercise, 4 hours post, 24 hours post, and 48 hours post) on 3 experimental trial days per participant (approximately 16 weeks total).
Menstrual Distress | From enrollment, through study completion, an average of 4 months.
  Description: Measure: Menstrual Distress Questionnaire (MEDI-Q). Objective: To examine the influence of the menstrual cycle on menstrual distress reporting. Time Frame: Assessed at 1 time point (baseline) on 3 experimental trial days per participant (approximately 16 weeks total)

OTHER OUTCOMES:
Cardiovascular Responses to Exercise | From enrollment, through study completion, an average of 4 months.
  Measure: Heart rate (beats per minute) recorded during exercise using a Polar H10 heart rate monitor. Objective: To measure the cardiovascular demand of resistance exercise and determine if it varies by menstrual phase.
  Time Frame: Continuously monitored during each exercise session on 3 experimental trial days (approximately 16 weeks total).
Exercise Enjoyment | From enrollment, through study completion, an average of 4 months.
  Measure: Physical Activity Enjoyment Scale (PACES; score range 18-126, higher scores = greater enjoyment). Objective: To evaluate whether menstrual cycle phases influence exercise enjoyment.
  Time Frame: Assessed immediately post-exercise on 3 experimental trial days (approximately 16 weeks total).
Rating of Perceived Exertion (RPE) | From enrollment, through study completion, an average of 4 months.
  Measure: Rating of Perceived Exertion (RPE; scale 6-20, higher = greater effort).
  Time Frame: Assessed after each exercise set and immediately post-exercise on 3 experimental trial days.
Repetitions in Reserve (RIR) | From enrollment, through study completion, an average of 4 months.
  Measure: Repetitions in Reserve (RIR; reps estimated to be left in reserve). Time Frame: Assessed after each exercise set on 3 experimental trial days.
Visual Analog Scale - Exercise Difficulty | From enrollment, through study completion, an average of 4 months.
  Measure: Visual Analog Scale (VAS; 0-100 mm, higher = more difficult). Time Frame: Assessed immediately post-exercise on 3 experimental trial days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Recruitment Website — https://healthprofessions.ucf.edu/research/studies/impact-of-the-menstrual-cycle-on-recovery-from-resistance-exercise/